CLINICAL TRIAL: NCT02245295
Title: Impact of Sedation Technique on the Diagnostic Accuracy of Endobronchial Ultrasound-guided Needle Aspiration (EBUS-TBNA)
Brief Title: The Role of Sedation Technique in EBUS-TBNA
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EBUSEDA1
Record Dates: First submitted 2014-09-15; First posted 2014-09-19 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Lung Cancer
Keywords: Bronchial endoscopy; ultrasound; EBUS; anesthesia; lung cancer; diagnosis including staging
MeSH Terms: conditions — Lung Neoplasms | interventions — Conscious Sedation; Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EBUS-TBNA: EBUS-TBNA for enlarged mediastinal/hilar lymph nodes
  Interventions: Procedure: Moderate Sedation for EBUS/TBNA; Procedure: General anesthesia for EBUS/TBNA

INTERVENTIONS:
Procedure: Moderate Sedation for EBUS/TBNA — EBUS-TBNA was performed by one of the pulmonologists in moderate sedation (D.F., M.K.).
Procedure: General anesthesia for EBUS/TBNA — EBUS-TBNA was performedin general anaesthesia by one of the thoracic surgeons (D.S., P.K.)

SUMMARY:
There is a paucity of data concerning the impact of the sedation technique used for endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) on diagnostic accuracy. The aim of this retrospective study is to compare diagnostic accuracy of EBUS-TBNA in deep and moderate sedation, and to investigate other possible determinants of diagnostic accuracy in three lymph node locations (mediastinal, subcarinal, and hilar).

The first consecutive patients at the University Hospital Zurich undergoing EBUS-TBNA for selective sampling in deep sedation are compared with the first consecutive patients in moderate sedation between 2006 and 2014. Diagnoses based on EBUS-TBNA were compared with those on surgical or radiological follow-up.

DETAILED DESCRIPTION:
Between September, 2007 and January 31, 2014, all consecutive patients who undergo EBUS-TBNA at the University Hospital Zurich for selective assessment of enlarged (≥ 1 cm by CT or ultrasound) or suspected (enhanced fluorodeoxyglucose (FDG) activity in PET/CT) lymph nodes were enrolled. Demographic and clinical data, procedural reports and cytological findings were collected from medical records. Computed tomography (CT) or PET/CT scans were prospectively reviewed to gather the size and standardized uptake value (SUV) of FDG of each sampled lymph node. The cytological findings obtained with EBUS-TBNA were verified by histological examination, if a surgical biopsy (mediastinoscopy, thoracoscopy, or thoracotomy) was carried out following EBUS-TBNA, or alternatively by clinical and radiological follow-up data.

ELIGIBILITY:
Inclusion Criteria:

* EBUS-TBNA

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with enlarged or suspicious mediastinal and/or hilar lymph nodes, in whom EBUS-TBNA is indicated
Sampling Method: Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1-6 months
  Sensitivity, negative predictive value

SECONDARY OUTCOMES:
Lymph node morphology | 1-6 months
  Impact of lymph node size on diagnostic accuracy
EBUS technique | 1-6 months
  Impact of EBUS technique (number of needle passes) on diagnostic accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, MD, Principal Investigator — Division of Pulmonology; Malcolm Kohler, Prof, Study Chair — Division of Pulmonology
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No